CLINICAL TRIAL: NCT00843414
Title: Immunological Characterization of Bronchoalveolar Cells in Normals
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Mark D. Wewers, MD, Associate Director of Pulmonary Research, Ohio State University
Other Study IDs: 1978H0059
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2011-04

CONDITIONS: Lung Disease
Keywords: Emphysema; Sarcoidosis; Interstitial Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases; Emphysema; Sarcoidosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood lung fluid (BAL)
Oversight: Data Monitoring Committee: No

SUMMARY:
To obtain the monocytes (white blood cells) from normal volunteers for the purpose of studying how proteins, fats, carbohydrates, as well as RNA and DNA for gene expression, relate to immunity. This information will be compared to other studies in patients with lung diseases such as Emphysema, Sarcoidosis, and Interstitial Pulmonary Fibrosis.

DETAILED DESCRIPTION:
To determine the functional capabilities of cells obtained from bronchoalveolar lavage fluid and peripheral blood monocytes from normal individuals. The ongoing objective varies from investigation to investigation but in general the investigational goals are to better understand the immune function of monocytes purified from normal volunteers. In some instances the emphasis will be upon comparing the specific immune function (e.g. ability to sense endotoxin and release a cytokine) from blood monocytes as compared to human alveolar macrophages. This comparison is not the only goal of the study, however. In many cases the immune function of the monocyte will be sufficient in and of itself as an investigational goal. In other cases the same is true of alveolar macrophage function.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 1232 (Actual)
Dates: Start 1978-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
comparing the specific immune function (e.g. ability to sense endotoxin and release a cytokine) from blood monocytes as compared to human alveolar macrophages | end of study

SECONDARY OUTCOMES:
Analysis of lung proteins present in BAL fluid | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Wewers, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States